CLINICAL TRIAL: NCT06293703
Title: Effect of Limb Length Ratio on Roux-en-Y Gastric Bypass Outcomes (CLIMB II Study)
Acronym: CLIMB II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salvador Navarrete (Other)
Responsible Party: Sponsor-Investigator, Salvador Navarrete, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-1228
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Morbid Obesity
Keywords: Bariatric surgery; Roux-n-Y gastric bypass; gastric bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, randomized controlled trial with a 1:1 recruitment allocation ratio coordinated at the Cleveland Clinic Foundation (CCF)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aRYGB (Experimental): BP and roux limb lengths measuring 30% and 15% respectively of patient's total small bowel length.
  Interventions: Procedure: Surgery
- sRYGB (Active Comparator): Standard fixed-length RYGB
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Biliopancreatic limb and roux limb lengths measuring 30 and 15% respectively of patient's total small bowel length in RYGB

SUMMARY:
The investigators propose a randomized controlled trial comparing BP and roux limb lengths measuring 30 and 15% respectively of patient's total small bowel length versus current standard practice using fixed lengths. The findings would provide further insight into feasibility of standardizing RYGB limb lengths and optimizing resultant weight loss and metabolic effects. The investigators hypothesize RYGB with ratio-adjusted limb lengths (aRYGB) will result in higher total weight loss and resolution of metabolic syndrome comorbidities, including diabetes, hyperlipidemia, and hypertension compared to standard fixed-length RYGB (sRYGB). The study will also utilize the Short Form Rand 36-Item Health Survey (SF36) to determine differences in postoperative quality of life metrics.

DETAILED DESCRIPTION:
This study will be a prospective, randomized controlled trial with a 1:1 recruitment allocation ratio. Patients will be randomized to Standard fixed-length RYGB (sRYGB) or ratio-adjusted limb lengths (aRYGB) once the total small bowel length (TSBL) is fully counted intraoperatively.

sRYGB will serve as the control group which will utilize BP and roux limb lengths of 100cm and 100cm, respectively. For the treatment group, aRYGB will incorporate a BP limb length measuring 30% and a roux limb of 15% of total small bowel length each.

Outcomes to be investigated:

Specific Aim 1: To determine significantly increased Total Weight Loss (TWL) after aRYGB compared to sRYGB in morbidly obese patients Given current understanding that weight loss after RYGB is mediated, at least in part, by a malabsorptive process, the investigators hypothesize that TWL will be greater after aRYGB versus sRYGB. As per standard of care at our institute, routine postoperative follow-up in the multidisciplinary Bariatric clinic will occur every 6 months (± 14 days) or more frequently as clinically indicated for the first two years postoperatively followed by yearly thereafter. Weight will be recorded in kilograms and a BMI will be calculated by the ratio of patient weight in kilograms over patient height in meters squared. Postoperative TWL will then be measured postoperatively at 6, 12, 24, 60 months from surgery.

Specific Aim 2: To compare rates of Diabetes Mellitus (DM) resolution between aRYGB Vs SRYGB by DM subgroup analysis Of the many metabolic changes that occur after bariatric surgery, one of the most salient effects include a rapid and effective resolution of DM. This has been extensively studied in context of various bariatric surgeries, including RYGB by our institution as previously described by the STAMPEDE trial. Significant reduction of HbA1C and improvement in insulin sensitivity was noted as early as six to 12 months postoperatively. As such, this study proposes measurement of the following two metrics at 6, 12, 24, 60 months postoperatively: 1) proportion of subjects achieving HbA1C less than or equal to 6.5%; and, 2) proportion of subjects able to wean and/or discontinue glycemic control medications.

Specific Aim 3: To investigate the relative postoperative efficacy of aRYGB compared to sRYGB on alleviating metabolic syndrome in morbid obesity Metabolic syndrome is a constellation of diagnoses including Hypertension (HTN) and Hyperlipidemia (HLD), which posit significant risk of medical comorbidities such as DM, coronary disease, and strokes. As such, addressing these conditions in morbidly obese patients confers a significant health benefit and decreases overall morbidity. This secondary outcome will be measured by comparing pre- versus postoperative serum lipid levels and proportion of patients requiring less antihypertensives 6, 12, 24, 60 months postoperatively.

Specific Aim 4: To investigate the presence of postoperative vitamin and nutritional deficiencies between the groups.

These secondary outcomes will be addressed comparing the vitamin levels between the groups at 6, 12, 24, 60 months postoperatively.

Additional outcomes proposed include evaluation of postoperative quality of life as captured by the Impact of Weight on Quality of Life-Lite-Clinical Trials (IWQOL-Lite-CT) survey as validated and effectively used in previous investigative bariatric studies. Responses will be tracked and obtained preoperatively and at various postoperative time points including Post-Operative Day (POD) 30 (± 15 days) and POD 365 (± 90 days). The investigators will furthermore track postoperative complications and adverse events, as measured by the Comprehensive Complications Index in addition to instances where additional bariatric surgical interventions are pursued.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients (defined by BMI between 40 and 60).
* Patient who understands and accepts the need for a long-term follow-up.
* Patient who agrees to be included in the study

Exclusion Criteria:

* individuals unable to understand and sign a written consent form
* patients with history of previous bariatric surgery procedures
* presence of a severe and evolutive life threatening pathology unrelated to obesity
* previous gastric or small bowel resection
* active cancer
* pregnancy or desired to be pregnant during the study
* mentally unbalanced patients under supervision or guardianship, patient unable to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2030-12-11 (Estimated)

PRIMARY OUTCOMES:
To determine change in TWL after aRYGB compared to sRYGB in morbidly obese patients | 6,12,24 and 60 months from surgery
  Measured in kilograms

SECONDARY OUTCOMES:
To compare rates of DM resolution between aRYGB Vs sRYGB by DM subgroup analysis | 6,12,24 and 60 months from surgery
  Measured by subjects achieving HbA1c less than or equal to 6.5% and subjects able to wean and/or discontinue glycemic control medications
To investigate postoperative efficacy rates of aRYGB compared to sRYGB on alleviating metabolic syndrome in morbid obesity | 6,12,24 and 60 months from surgery
  Measured by a change in serum lipid levels and subjects requiring less antihypertensives
To investigate the presence of postoperative vitamin and nutritional deficiencies between the groups. | 6,12,24 and 60 months from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Navarrete, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided